CLINICAL TRIAL: NCT05177445
Title: Efficacy and Safety of Phototherapy in the Treatment of Loss of Smell Post Acute Infection of Coronavirus 19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Respiralab (Other)
Responsible Party: Principal Investigator, Ivan Cherrez Ojeda, Research Professor of Allergy, Immunology and Pulmonology, Respiralab
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HCK-RNLTA-19-0007
Record Dates: First submitted 2021-10-15; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Smell Disorders
Keywords: Anosmia; Hyposmia; Coronavirus; Smell Disorders; Phototherapy
MeSH Terms: conditions — Olfaction Disorders; Anosmia; Coronavirus Infections | interventions — Phototherapy; Adrenal Cortex Hormones; Olfactory Training

STUDY DESIGN:
Intervention Model Description: Interventional study, single blinded, convenience sampling.
Who Masked: Participant
Masking Description: Patients will receive information about both treatments, but won't have knowledge about which treatment is applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group with phototherapy (Experimental): Patients that present loss of smell 4 weeks after their coronavirus-19 infection and that have had a real-time polymerase chain reaction (reverse transcriptase polymerase chain reaction ) positive for coronavirus-19 will receive the phototherapy intervention. It consists of the introduction of the nasal probe of the phototherapy device in the nasal cavity of the patient. A mixture of ultraviolet light A, ultraviolet light B and red light will be applied between 2 and 3 minutes. The patient will receive a maximum of 10 interventions. Furthermore both oral corticosteroids (prednisone 40mg) and olfactory training will be applied, in the intervals of daily for 10 days and daily for the duration of the study respectively.
  Interventions: Combination Product: Phototherapy
- Intervention group (corticosteroids + OT) without Phototherapy (Active Comparator): Patients that present loss of smell 4 weeks after their coronavirus-19 infection and that have had a real-time polymerase chain reaction (reverse transcriptase polymerase chain reaction )and both oral corticosteroids (prednisone 40mg) and olfactory training will be applied, in the intervals of daily for 10 days and daily for the duration of the study respectively.
  Interventions: Combination Product: OT+Corticosteroids

INTERVENTIONS:
Combination Product: Phototherapy — Prior to the beginning of the procedure the patient will be administered a nasal decongestant. Second to this, the patient will be advised to blow his/her nose. This step allows the physician a better view and allows the light exposure to reach the majority of the nasal mucosa(9).
  To start the intervention the physician will introduce the phototherapy device inside the patient's nasal cavity as the patient sits in an upright condition. As the procedure is ongoing the physician will slightly rotate the device in order to minimize dryness and to irradiate all the nasal cavity. After the intervention the patient will be administered an emollient/moisturizing drug to further hydrate the nasal mucosa(9).
  The intervention will have a crescent duration, the first one will be only two minutes and the following ones will increase 15 seconds each until a plateau is reached at 3 minutes in the 5th intervention.
  Other Names: Corticosteroids; Olfactory training
  Arms: Intervention group with phototherapy
Combination Product: OT+Corticosteroids — Patients that present loss of smell 4 weeks after their coronavirus-19 infection and that have had a real-time polymerase chain reaction (reverse transcriptase polymerase chain reaction )and both oral corticosteroids (prednisone 40mg) and olfactory training will be applied, in the intervals of daily for 10 days and daily for the duration of the study respectively.
  Other Names: Corticosteroid; Olfactory training
  Arms: Intervention group (corticosteroids + OT) without Phototherapy

SUMMARY:
The aim of this study is to assess whether the use of a therapy combining olfactory training, corticoids, and phototherapy improves the PROMS compared to the use of olfactory training and corticosteroids only. To accomplish this goal the study will consist of 40 participants. The participants must present olfactory dysfunction for at least 4 weeks after a coronavirus-19 infection. Furthermore, to be eligible each participant will need a polymerase chain reaction test with positive results for coronavirus-19.

DETAILED DESCRIPTION:
Standard Operating Procedures: Patients attending consult and calls for follow-up.

Plan for missing data: Missing data will be managed with statistical tests.

Statistical analysis: Categorical variables, whenever dichotomous or nominal, will be reported as frequencies and percentages. Normality will be assessed by the Kolmogorov Smirnov test. Descriptive statistics will be reported as mean (standard deviation) or median (interquartile range). To analyze the correlation between quantitative variables, the parametric Pearson test or the nonparametric Spearman's test will be used, subjected to their distribution. Differences between Diffusing capacity for carbon monoxide groups will be analyzed for statistical significance by the chi-square test for categorical variables and by a two-sample t-test or Wilcoxon rank-sum test for continuous variables as applicable. Statistical significance will be set at a P-value less than 0.05. Analyses will be performed using Statistical Package for the Social Sciences (V. 22.0) software.

ELIGIBILITY:
Inclusion Criteria:

* Positive coronavirus polymerase chain reaction patients who experience loss of smell for more than 4 weeks after symptoms begin will be included in the study but at time of the trial with a negative result from a polymerase chain reaction.
* Patients older than18 years.

Exclusion Criteria:

* Patients younger than 18 years.
* Pregnancy.
* Patients who do not have a positive real-time polymerase chain reaction for Coronavirus
* Patients who have contraindications for corticosteroid therapy such as:

  1. Pregnant patients
  2. Immunosuppressed
  3. Patients with peptic ulcer
  4. Diabetics
  5. Patients with glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change of Loss of Smell in Visual Analog Scale (VAS) | It will be assessed through the study completion, an average of 15 weeks.
  The Visual Analog Scale (VAS) scale is able to determine the grade of loss of smell. From 1 to 10, being 1 the minimum and 10 the maximum grade of loss of smell.
Changes in the Threshold Discrimination Identification (TDI) score | It will be assessed through the study completion, an average of 15 weeks.
  The Threshold Discrimination Identification score (TDI) is used when the patient undergoes olfactory training, it is comprised by 3 tests: the threshold, discrimination, and identification. Each result is interpreted according to 4 age groups.
  The test is accomplished by having the patient sniff at a felt pen which has been impregnated with 4ml of odorant fluid dissolved in propylene glycol. TDI scores defined functional anosmia as a TDI score <16,5, normosmia as a TDI score >30.5 and hyposmia as a score between these two values.
Changes of olfactory dysfunction in the Self-reported mini olfactory questionnaire (Self-MOQ) | It will be assessed through the study completion, an average of 15 weeks.
  The Self-reported mini olfactory questionnaire (Self-MOQ) is a simple, reliable and valid questionnaire to screen olfactory dysfunction in clinical practice. For the sample in the current study, the optimal scores will be 3.5, 4.5, and 3.5 for distinguishing normosmic from hyposmic/ anosmic patients, anosmic patients, and hyposmic patients, respectively.

SECONDARY OUTCOMES:
Changes in Anxiety and depression in the Hospital Anxiety and Depression Scale(HADS) | It will be assessed through the study completion, an average of 15 weeks.
  The Hospital Anxiety and Depression Scale (HADS) allows for the assessment of both anxiety and depression as it has been seen that both can be present at the same time. This scale focuses on non-physical symptoms so that it can be used to diagnose depression in people with significant physical illness.
  The questionnaire comprises seven questions for both anxiety and depression, and should take around 2-5min to complete. A score between 8 and 10 is considered as mild, if it is between 11 and 14 it is considered moderate and if it exceeds 15 it is considered severe.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel I Cherrez Ojeda, MD. MsC., Principal Investigator — RESPIRALAB RESEARCH GROUP
Locations (1):
- Respiralab Research Group, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cingi C, Yaz A, Cakli H, Ozudogru E, Kecik C, Bal C. The effects of phototherapy on quality of life in allergic rhinitis cases. Eur Arch Otorhinolaryngol. 2009 Dec;266(12):1903-8. doi: 10.1007/s00405-009-1048-y. Epub 2009 Jul 22. PMID 19626333
- [Background] Beissert S, Schwarz T. Role of immunomodulation in diseases responsive to phototherapy. Methods. 2002 Sep;28(1):138-44. doi: 10.1016/s1046-2023(02)00217-7. PMID 12231198
- [Background] Matz H. UV light and its interaction with cutaneous receptors. Dermatol Clin. 2007 Oct;25(4):633-41, x. doi: 10.1016/j.det.2007.06.006. PMID 17903622
- [Background] Le Bon SD, Konopnicki D, Pisarski N, Prunier L, Lechien JR, Horoi M. Efficacy and safety of oral corticosteroids and olfactory training in the management of COVID-19-related loss of smell. Eur Arch Otorhinolaryngol. 2021 Aug;278(8):3113-3117. doi: 10.1007/s00405-020-06520-8. Epub 2021 Jan 9. PMID 33423106
- [Background] Brehmer D. Endonasal phototherapy with Rhinolight for the treatment of allergic rhinitis. Expert Rev Med Devices. 2010 Jan;7(1):21-6. doi: 10.1586/erd.09.56. PMID 20021238
- [Background] Novak Z, Berces A, Ronto G, Pallinger E, Dobozy A, Kemeny L. Efficacy of different UV-emitting light sources in the induction of T-cell apoptosis. Photochem Photobiol. 2004 May;79(5):434-9. doi: 10.1562/ra-003r.1. PMID 15191052
- [Background] O'Byrne L, Webster KE, MacKeith S, Philpott C, Hopkins C, Burton MJ. Interventions for the treatment of persistent post-COVID-19 olfactory dysfunction. Cochrane Database Syst Rev. 2021 Jul 22;7(7):CD013876. doi: 10.1002/14651858.CD013876.pub2. PMID 34291813